CLINICAL TRIAL: NCT01900652
Title: A Randomized, Open-Label Phase 2 Study Evaluating LY2875358 Plus Erlotinib and LY2875358 Monotherapy in MET Diagnostic Positive NSCLC Patients With Acquired Resistance to Erlotinib
Brief Title: A Study of Emibetuzumab in Non Small Cell Lung Cancer (NSCLC) Participants
Acronym: Chime
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14208; I4C-MC-JTBC (Other: Eli Lilly and Company)
Record Dates: First submitted 2013-07-12; First posted 2013-07-16 (Estimated); Results first posted 2018-06-25 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — emibetuzumab; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A: Emibetuzumab plus Erlotinib (Experimental): 750 milligram (mg) Emibetuzumab flat dose given as a 1.5 hour intravenous (IV) infusion on Days 1 and 15 of a 28-day cycle and Erlotinib 150 mg given orally once daily on a 28-day cycle.
  Interventions: Drug: Emibetuzumab; Drug: Erlotinib
- Arm B: Emibetuzumab (Experimental): 750 mg Emibetuzumab flat dose given as a 1.5-hour IV infusion on Days 1 and 15 of a 28-day cycle.
  Interventions: Drug: Emibetuzumab

INTERVENTIONS:
Drug: Emibetuzumab — Administered IV
  Other Names: LY2875358
Drug: Erlotinib — Administered Orally
  Arms: Arm A: Emibetuzumab plus Erlotinib

SUMMARY:
The primary purpose of this study is to evaluate the efficacy of the study drug known as LY2875358, administered alone or in combination with a second drug named Erlotinib, in participants affected by a defined type of lung cancer (MET biomarker diagnostic positive Non-Small-Cell Lung Cancer) that experienced a disease progression during the most recent treatment with Erlotinib.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of metastatic Stage IV NSCLC
* At least 1 measurable extra-central nervous system (CNS) lesion
* Documented radiographic progression while on continuous treatment with erlotinib monotherapy
* Objective clinical benefit from erlotinib treatment as defined by either documented partial or complete response or stable disease ≥6 months or, if most recent erlotinib treatment has been initiated based on documented epidermal growth factor receptor mutation (EGFRmt) status, at least 12 weeks stable disease
* Determined to be MET diagnostic positive (+)
* Availability of a tumor sample post-erlotinib progression
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2
* Have adequate organ function

Exclusion Criteria:

* Are currently enrolled in, or discontinued within the last 30 days from, a clinical trial involving an investigational product or non-approved use of a drug or device
* Have previously been treated with LY2875358 or any other MET-targeting experimental therapeutic
* Have a serious concomitant systemic disorder or significant cardiac disease
* Have interstitial pneumonia or interstitial fibrosis of the lung or have pleural effusion, pericardial fluids or ascites, requiring drainage every other week or more frequently
* Have a history of another malignancy except for basal or squamous cell skin cancer and/or in situ carcinoma of the cervix, or other solid tumors treated curatively and without evidence of recurrence for at least 3 years prior to the study
* Have major surgery less than 2 weeks prior initiation of study treatment therapy
* Pregnant or lactating women
* Have symptomatic CNS metastasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2013-08; Primary Completion 2015-02 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (59):
- United States (32):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California - San Diego, La Jolla, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Los Angeles, California
  - University of California, Davis - Health Systems, Sacramento, California
  - UCLA, Santa Monica, California
  - University of Colorado Health Sciences Center, Aurora, Colorado
  - Georgetown University Medical Center IRB, Washington D.C., District of Columbia
  - Florida Cancer Specialists, Fort Myers, Florida
  - Florida Cancer Specialists, St. Petersburg, Florida
  - H Lee Moffitt Cancer Center, Tampa, Florida
  - Northeast Georgia Cancer Care, LLC, Athens, Georgia
  - Emory University, Atlanta, Georgia
  - University of Iowa Hospital, Iowa City, Iowa
  - University of Kansas Medical Center, Westwood, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Washington University Medical Center, St Louis, Missouri
  - Billings Clinic Research Center, Billings, Montana
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Columbia University, New York, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Oncology Hematology Care Inc, Cincinnati, Ohio
  - Portland VA Medical Center, Portland, Oregon
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Tennessee Oncology PLLC, Chattanooga, Tennessee
  - The West Clinic, Memphis, Tennessee
  - Tennessee Oncology PLLC, Nashville, Tennessee
  - MS Center at Evergreen, Kirkland, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Group Health, Seattle, Washington
  - Multicare Health System, Tacoma, Washington
- Belgium (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aalst
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ghent
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mechelen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Roeselare
- France (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Montpellier
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toulouse
- Germany (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heidelberg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ulm
- Israel (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beersheba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jerusalem
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kfar Saba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Petah Tikva
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tel Litwinsky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ẕerifin
- Italy (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Milan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orbassano
- Netherlands (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Amsterdam
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Breda
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul, South Korea
- Spain (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Badalona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pamplona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Valencia
- United Kingdom (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bristol, Avon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London, Greater London
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Southampton, Hants
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wythenshawe, Manchester
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Headington, Oxford

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm B: Emibetuzumab 750mg: 750 mg Emibetuzumab flat dose given as a 1.5-hour IV infusion on Days 1 and 15 of a 28-day cycle.
Period: Overall Study
Arm/Group | Arm A: Emibetuzumab Plus Erlotinib | Arm B: Emibetuzumab 750mg
Started | 83 | 28
Post-Erlotinib Progression Tumor Sample | 66 | 23
Completed | 75 | 25
Not Completed | 8 | 3
Not completed — Progressive Disease | 1 | 0
Not completed — Consent withdrawn by subject | 1 | 1
Not completed — Death | 3 | 0
Not completed — Adverse Event | 2 | 1
Not completed — Physician Decision | 1 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least one dose of study drug.
Groups:
- Arm A: Emibetuzumab Plus Erlotinib: 750 milligram (mg) Emibetuzumab (LY2875358) flat dose given as a 1.5 hour intravenous (IV) infusion on Days 1 and 15 of a 28-day cycle and Erlotinib 150 mg given orally once daily on a 28-day cycle.
- Total: Total of all reporting groups
Arm/Group | Arm A: Emibetuzumab Plus Erlotinib | Arm B: Emibetuzumab | Total
Number analyzed (Participants) | 83 | 28 | 111
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.2 (10.8) | 60.9 (12.0) | 63.3 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 20 | 75
  Male | 28 | 8 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 0 | 4
  Not Hispanic or Latino | 70 | 21 | 91
  Unknown or Not Reported | 9 | 7 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 10 | 3 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 0 | 4
  White | 64 | 23 | 87
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 4 | 2 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  Netherlands | 5 | 5 | 10
  Belgium | 9 | 0 | 9
  United States | 32 | 9 | 41
  South Korea | 3 | 3 | 6
  Italy | 3 | 0 | 3
  United Kingdom | 6 | 3 | 9
  Israel | 7 | 4 | 11
  France | 5 | 2 | 7
  Germany | 4 | 1 | 5
  Spain | 9 | 1 | 10
ECOG Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) classifies participants according to their functional impairment. Scores range from 0 (Fully Active) to 5 (Death). 0 - Fully Active. 1 - Ambulatory, Restricted Strenuous Activity. 2 - Ambulatory, No Work Activities. 3 - Partially Confined to Bed, Limited Self Care. 4 - Completely Disabled. 5 - Death.
  Participants
    ECOG 0 | 18 | 9 | 27
    ECOG 1 | 60 | 17 | 77
    ECOG 2 | 5 | 2 | 7
Pathological Diagnosis [Count of Participants; unit: Participants]
  Lung Adenocarcinoma | 77 | 22 | 99
  Squamous Cell Carcinoma | 3 | 1 | 4
  Large Cell Carcinoma | 0 | 1 | 1
  Other Subtypes of Lung Cancer | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Complete Response (CR) or Partial Response (PR) (Overall Response Rate [ORR])
Description: ORR is confirmed best overall tumor response of CR or PR. According to RECIST v1.1, CR was defined as the disappearance of all target and non-target lesions; PR defined as a >30% decrease in the sum of the longest diameters (LD) of the target lesions, taking as reference the baseline sum of the LD. Percentage of participants was calculated as: (total number of participants with CR or PR from start of the treatment until disease progression or recurrence)/total number of participants treated) * 100.
Time Frame: Baseline to Objective Disease Progression or Start of New Anticancer Therapy (Up to 15 Months)
Population: All participants who are MET diagnostic positive based on the results of their post-erlotinib progression tumor sample and resistance to erlotinib.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- MET-High Analysis Population (Emibetuzumab + Erlotinib): Participants in the Emibetuzumab + Erlotinib treatment arm with MET-High expression status based on their post-erlotinib progression NSCLC tumor sample.
- MET-High Analysis Population (Emibetuzumab): Participants in the Emibetuzumab treatment arm with MET-High expression status based on their post- erlotinib progression NSCLC tumor sample.
Arm/Group | Arm A: Emibetuzumab Plus Erlotinib | Arm B: Emibetuzumab | MET-High Analysis Population (Emibetuzumab + Erlotinib) | MET-High Analysis Population (Emibetuzumab)
Number analyzed (Participants) | 66 | 23 | 53 | 21
percentage of participants | 3.0 [0.4 to 10.5] | 4.3 [0.1 to 21.9] | 3.8 [0.5 to 13.0] | 4.8 [0.1 to 23.8]

2. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS defined as date of randomization until the date of objectively determined progression defined by Response Evaluation Criteria in Solid Tumors criteria or death from any cause, whichever is first.
  Progressive disease (PD) defined as ≥20% increase in sum of diameter of target lesion with the sum demonstrating an increase of ≥5 mm; appearance of ≥1 new lesions or unequivocal progression of non- target lesions. Participants with no baseline disease assessment were censored at randomization date, regardless of whether or not objectively determined PD or death was observed; participants not known to have died or to have objective progression as of data inclusion cutoff were censored at last post baseline radiological assessment date or randomization date, if there was no post baseline radiological assessment.
Time Frame: Baseline to Objective Disease Progression or Death (Up to 24 Months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Emibetuzumab Plus Erlotinib | Arm B: Emibetuzumab
Number analyzed (Participants) | 66 | 23
Months | 3.3 [1.7 to 4.2] | 1.6 [1.2 to 3.1]

3. Secondary Outcome: Time to Progressive Disease
Time Frame: Baseline to Objective Disease Progression (Up to 24 Months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Emibetuzumab Plus Erlotinib | Arm B: Emibetuzumab
Number analyzed (Participants) | 66 | 23
months | 3.8 [2.7 to 4.7] | 1.6 [1.4 to 3.1]

4. Secondary Outcome: Change in Tumor Size (CTS)
Description: Zero participants analyzed. CTS data was not collected for analysis due to N=0 CR and N=3 PR.
Time Frame: Baseline to Measurement with Smallest Tumor Size (Up to 24 Months)
Population: Zero participants analyzed.CTS data was not collected for analysis due to N=0 CR and N=3 PR.
Groups:
- Arm B: LY2875358: 750 mg Emibetuzumab flat dose given as a 1.5-hour IV infusion on Days 1 and 15 of a 28-day cycle.
Arm/Group | Arm A: Emibetuzumab Plus Erlotinib | Arm B: LY2875358
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Secondary: Percentage of Participants Who Achieved Best Overall Disease Response of CR, PR or Stable Disease (SD) [Disease Control Rate (DCR)]
Description: Participants achieved disease control if they had a best overall response of PR, CR or SD. According to RECIST v1.1, CR was the disappearance of all non-nodal target lesions, with the short axes of any target lymph node reduced to <10 mm, the disappearance of all nontarget lesions, and the normalization of tumor marker levels (if tumor markers were initially above the upper limit of normal [ULN]); PR was defined as at least a 30% decrease in the sum of the diameters of target lesions (including the short axes of any target lymph node), taking as reference the baseline sum diameter. SD was neither sufficient shrinkage to qualify as PR nor sufficient increase to qualify as PD, taking as reference the smallest sum diameter since treatment started. The percentage of participants who achieved disease control equals (number of participants with CR, PR, or SD)/(number of participants assessed)*100.
Time Frame: Baseline to Objective Disease Progression or Participant Stops Study (Up to 24 Months)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: Emibetuzumab Plus Erlotinib | Arm B: Emibetuzumab | MET-High Analysis Population (Emibetuzumab + Erlotinib) | MET-High Analysis Population (Emibetuzumab)
Number analyzed (Participants) | 66 | 23 | 53 | 21
percentage of participants | 50 [37.4 to 62.6] | 26.1 [10.2 to 48.4] | 47.2 [33.3 to 61.4] | 28.6 [11.3 to 52.2]

6. Secondary Outcome: Duration of Response (DoR)
Description: Zero participants analyzed. Duration of Response for CR and PR data was not collected for analysis due to N=0 CR and N=3 PR.
Time Frame: Date of CR or PR to Date of Objective Disease Progression or Death Due to Any Cause (Up to 24 Months)
Population: Zero participants analyzed. Duration of Response for CR and PR data was not collected for analysis due to N=0 CR and N=3 PR.
Arm/Group | Arm A: Emibetuzumab Plus Erlotinib | Arm B: Emibetuzumab
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as duration from the date of study enrollment to the date of death from any cause. Participants not known to have died as of the data inclusion cut-off date were censored at the date of last contact. The last contact for participants in post-discontinuation was the last date participant was known to be alive.
Time Frame: Baseline to Death Due to Any Cause (Up to 24 Months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Emibetuzumab Plus Erlotinib | Arm B: Emibetuzumab
Number analyzed (Participants) | 66 | 23
Months | 9.2 [6.7 to 12.0] | 8.2 [3.7 to 12.6]

8. Secondary Outcome: Change From Baseline in European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaires C30 (QLQ-C30)
Description: EORTC QLQ-C30 v3.0 is a self-administered questionnaire with multidimensional scales that measures 5 functional domains (physical, role, cognitive, emotional, and social), global health status, and symptom scales of fatigue, pain, nausea and vomiting, dyspnea, loss of appetite, insomnia, constipation and diarrhea, and financial difficulties. A linear transformation is applied to standardize the raw scores to range between 0 and 100 per developer guidelines. For functional domains and global health status, higher scores represent a better level of functioning. For symptoms scales, higher scores represented a greater degree of symptoms.
Time Frame: Baseline, Objective Disease Progression or Participants Stops Study (Up to 24 Months)
Population: All randomized participants with EORTC QLQ-C30 values at baseline.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- MET-High Analysis Population: Participants with MET-High expression status based on their post-erlotinib progression NSCLC tumor sample.
Arm/Group | Arm A: Emibetuzumab Plus Erlotinib | Arm B: Emibetuzumab | MET-High Analysis Population
Number analyzed (Participants) | 83 | 28 | 74
units on a scale
  QoL | -4.0 (18.3) | -21.9 (18.9) | -10.2 (22.3)
  Physical | -11.4 (25.8) | -22.9 (30.2) | -19.0 (27.4)
  Role | -7.7 (42.0) | -35.4 (35.0) | -21.0 (39.3)
  Emotional | 1.7 (29.9) | -13.5 (19.9) | -6.1 (29.7)
  Cognitive | -3.3 (31.2) | -10.4 (25.1) | -9.8 (29.4)
  Social | -12.5 (29.6) | -16.7 (39.8) | -19.8 (29.2)
  Fatigue | 8.5 (23.6) | 31.9 (33.8) | 16.9 (30.7)
  Nausea/vomiting | -1.3 (31.2) | 0 (0) | 0.7 (39.1)
  Pain | 1.9 (26.0) | 14.6 (24.3) | 2.2 (28.6)
  Dyspnea | 9.0 (32.1) | 29.2 (37.5) | 14.5 (38.7)
  Insomnia | -14.1 (39.1) | -16.7 (23.6) | -15.9 (43.7)
  Appetite Loss | 6.4 (36.5) | 29.2 (41.5) | 15.9 (42.5)
  Constipation | 3.8 (31.7) | 33.3 (50.4) | 17.4 (38.8)
  Diarrhea | -5.3 (41.6) | 4.2 (48.6) | -1.5 (43.0)
  Finance | -6.7 (23.6) | 8.3 (42.7) | 3.0 (30.7)

9. Secondary Outcome: Change From Baseline in EORTC Quality of Life Questionnaires Lung Cancer 13 (QLQ-LC13)
Description: The EORTC lung module QLQ-LC13 comprises 13 items consisting of one multi-item scale to assess dyspnea and a series of single-item measures assessing pain, coughing, sore mouth, dysphagia, peripheral neuropathy, alopecia, and hemoptysis. A linear transformation is applied to standardize the raw scores to range between 0 and 100 per developer guidelines. The higher scores represent a greater degree of symptoms.
Time Frame: Baseline, Objective Disease Progression or Participants Stops Study (Up to 24 Months)
Population: All randomized participants with EORTC QLQ-LC13 values at baseline.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm A: Emibetuzumab Plus Erlotinib | Arm B: Emibetuzumab | MET-High Analysis Population
Number analyzed (Participants) | 83 | 28 | 74
units on a scale
  Coughing | 14.1 (35.5) | 16.7 (35.0) | 17.5 (35.9)
  Hemoptysis | 2.6 (9.1) | 0 (0) | 3.2 (10.0)
  Sore Mouth | 7.7 (25.5) | 5.6 (13.6) | 12.7 (22.3)
  Dysphagia | 7.7 (25.5) | 5.6 (13.6) | 9.5 (26.1)
  Peripheral Neuropathy | -5.1 (22.5) | 5.6 (13.6) | -4.8 (21.8)
  Alopecia | -5.3 (34.3) | 0 (0) | 4.8 (19.1)
  Pain in Chest | -1.3 (11.7) | 5.6 (13.6) | 1.7 (13.1)
  Pain in Shoulder or Arm | -2.6 (28.2) | 0 (0) | 3.2 (25.6)
  Pain in Other Parts | 8.0 (30.9) | 16.7 (45.9) | 3.3 (32.3)

10. Secondary Outcome: Change From Baseline in EuroQol 5-Dimensional Scale (EQ-5D)
Description: The EQ-5D is a generic, multidimensional, health status instrument. The profile allows participants to rate their health state in 5 health domains: mobility, self-care, usual activities, pain/discomfort, and mood using a 3-level scale (no problem, some problems, and major problems). These combinations of attributes were converted into a weighted health-state Index Score according to the United Kingdom (UK) population-based algorithm. The possible values for the Index Score ranged from -0.59 (severe problems in all 5 dimensions) to 1.0 (no problem in any dimension). A negative change indicated a worsening of the participant's health status.
  Additionally, participants will indicate their current health status by marking on a continuum ranging from 100 (best imaginable health state) to 0 (worst imaginable health state).
Time Frame: Baseline, Objective Disease Progression or Participants Stops Study (Up to 24 Months)
Population: All randomized participants with EQ-5D values at baseline.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm A: Emibetuzumab Plus Erlotinib | Arm B: Emibetuzumab | MET-High Analysis Population
Number analyzed (Participants) | 78 | 22 | 64
units on a scale
  Index Score | -0.1 (0.3) | -0.2 (0.3) | -0.1 (0.3)
  Visual Analog Scale | -8.3 (18.0) | -12.5 (21.7) | -11.8 (19.4)

11. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration (AUC) of Emibetuzumab
Description: AUC(0-tlast) = area under the concentration versus time curve from time zero through the last quantifiable sample.
Time Frame: Cycle1 Day 1 (C1 D1): Pre-dose and End of infusion; C1 D8: Pre-dose; C1 D15, C2 D1, C2 D15, C3 D1, C3 D15, C4 D1, C4 D15: Pre-dose and End of Infusion
Population: All participants who received Emibetuzumab on Cycle 1, Day 1, and contributed samples for analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram*hour/milliliter (ug*hr/mL)
Groups:
- Emibetuzumab: All participants who received Emibetuzumab on Cycle 1, Day 1, and contributed samples for analysis.
Arm/Group | Emibetuzumab
Number analyzed (Participants) | 19
Microgram*hour/milliliter (ug*hr/mL) | 31400 (75)

12. Secondary Outcome: Number of Participants With Anti-Emibetuzumab Antibody (ADA) Response
Time Frame: Baseline through 30-Day Follow-Up (Up to 24 Months)
Population: All participants who received at least one dose of study drug and have sufficient Anti-Emibetuzumab Antibody sample for the analysis.
Measure: Number; unit: participants
Arm/Group | Arm A: Emibetuzumab Plus Erlotinib | Arm B: Emibetuzumab
Number analyzed (Participants) | 44 | 17
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Through study completion and the 30-day post-discontinuation follow-up period (up to 24 months).
Arm/Group | Arm A: Emibetuzumab Plus Erlotinib | Arm B: Emibetuzumab
All-Cause Mortality (participants affected / at risk) | 0/83 | 0/28
Serious Adverse Events (participants affected / at risk) | 36/83 | 11/28
Other Adverse Events (participants affected / at risk) | 82/83 | 28/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Emibetuzumab Plus Erlotinib (N=83) | Arm B: Emibetuzumab (N=28)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (4) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 3 (3) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 1 (1)
Pain (General disorders) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Rash pustular (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 1 (2)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Tracheobronchitis (Infections and infestations) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 1 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 2 (3)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Emibetuzumab Plus Erlotinib (N=83) | Arm B: Emibetuzumab (N=28)
Anaemia (Blood and lymphatic system disorders) | 11 (16) | 3 (3)
Tachycardia (Cardiac disorders) | 1 (1) | 2 (2)
Lacrimation increased (Eye disorders) | 0 (0) | 2 (2)
Vision blurred (Eye disorders) | 1 (1) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 3 (5)
Constipation (Gastrointestinal disorders) | 18 (21) | 8 (8)
Diarrhoea (Gastrointestinal disorders) | 21 (36) | 7 (9)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 (6) | 2 (2)
Nausea (Gastrointestinal disorders) | 27 (32) | 7 (7)
Stomatitis (Gastrointestinal disorders) | 9 (11) | 2 (2)
Vomiting (Gastrointestinal disorders) | 16 (24) | 6 (8)
Asthenia (General disorders) | 9 (19) | 5 (5)
Axillary pain (General disorders) | 1 (1) | 3 (3)
Chills (General disorders) | 2 (2) | 2 (2)
Fatigue (General disorders) | 40 (59) | 11 (15)
Non-cardiac chest pain (General disorders) | 5 (5) | 2 (2)
Oedema peripheral (General disorders) | 30 (42) | 9 (15)
Pain (General disorders) | 0 (0) | 2 (3)
Pyrexia (General disorders) | 4 (5) | 4 (4)
Paronychia (Infections and infestations) | 11 (18) | 0 (0)
Urinary tract infection (Infections and infestations) | 6 (10) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Activated partial thromboplastin time prolonged (Investigations) | 1 (2) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 6 (8) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 6 (7) | 1 (1)
Prothrombin time prolonged (Investigations) | 0 (0) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 25 (27) | 4 (4)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 13 (25) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 7 (7) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (13) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (8) | 1 (3)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7 (7) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (3) | 3 (3)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (9) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (10) | 4 (4)
Dizziness (Nervous system disorders) | 5 (5) | 1 (1)
Headache (Nervous system disorders) | 5 (5) | 3 (4)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (3)
Insomnia (Psychiatric disorders) | 7 (7) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 17 (21) | 8 (8)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 22 (30) | 8 (11)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (8) | 3 (3)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 15 (23) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 8 (8) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 9 (24) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 (8) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 7 (7) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days